CLINICAL TRIAL: NCT04822493
Title: Improving Pain Perceptions After Initiating a Delivery Application
Acronym: iPANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00099027
Record Dates: First submitted 2020-09-11; First posted 2021-03-30 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Pain; Pain
Keywords: Pain perception; Postpartum; Counseling aid; ERAS; Postpartum pain; Pain expectations
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: The investigators plan to use block randomization with stratification. The randomization schedule will have 1:1 allocation with a fixed block size of 4. To ensure equivalent numbers for planned cesarean and planned vaginal deliveries, patients will be stratified based on expected mode of delivery.
  Randomization will occur at the time of enrollment. A computer-generated randomization scheme has been developed within the mobile application. When the participant is assigned a study number, the application with randomly assign them to the study or control group, based on the scheme described above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling Aid (Experimental): A. Complete the demographic questionnaire, the survey questions, and then complete the counseling aid. Receive standard counseling as part of routine prenatal care.
  B. Prior to discharge after delivery, study personnel will administer the postpartum questionnaire via a mobile tablet. The questionnaire is programmed into the study application.
  Interventions: Other: Counseling Aid
- Standard Care (No Intervention): A. Complete the demographic questionnaire and survey questions without watching the educational video. Receive standard counseling as part of routine prenatal care.
  B. Prior to discharge after delivery, study personnel will administer the postpartum questionnaire via a mobile tablet. The questionnaire is programmed into the study application.

INTERVENTIONS:
Other: Counseling Aid — Women will watch an educational video regarding expectations for delivery and postpartum care in addition to receiving standard care and counseling.
  Arms: Counseling Aid

SUMMARY:
The investigators of this study have developed a standardized counseling aid using an electronic mobile device to help women learn about what to expect during labor and subsequent vaginal delivery or cesarean delivery, specifically regarding pain expectations. Half of women will complete the counseling aid and the other half will receive standard counseling and care. The study aims to determine if the counseling aid improves patient satisfaction and perception of pain control.

DETAILED DESCRIPTION:
A. Objective To compare perception of postpartum pain and patient satisfaction between women who receive routine obstetric care to those who receive routine obstetric care and complete a standardized counseling aid antepartum.

B. Background Enhanced Recovery After Surgery (ERAS) is a standardized, evidenced-based method for the perioperative management of surgical patients. ERAS protocols have been well studied in several surgical specialties, including gynecologic oncology and benign gynecology, and have been shown to reduce hospital length of stay and costs without increasing rates of complications or readmission.

The use of ERAS in obstetrics is also growing. Recent studies have shown that an enhanced recovery pathway after cesarean delivery can decrease hospital stay and cost and reduce opioid use. Guidelines have been developed for evidence-based recommendations for preoperative, intraoperative and postoperative phases of care.

An important component of any ERAS protocol is pre-operative counseling. Postoperative pain management starts with counseling prior to surgery. Guidelines suggest that preoperative counseling should include patient-centered education on the options for management of pain. This process also allows an opportunity to engage patients in the decision making process. Previous studies have shown that counseling on pain expectations can improve patient outcomes.

The aim of our study is to develop a standardized antepartum counseling aid and improve postpartum pain perceptions and patient experience.

C. Study Methodology

1. Study Design The study is a randomized control trial. Patients will be assigned 1:1 to the study group and control group.
2. Comparison Groups:

1: Group 1:

* Study Group: Women will watch an educational video regarding expectations for delivery and postpartum care in addition to receiving standard care and counseling.

  2: Group 2:
* Control Group: Women will receive standard care and counseling.

  3. Procedures:

Identification of Potentially Eligible Patients

1. Potentially eligible patients will be identified through screening of clinic patients at time of routine prenatal visit at the Prisma Health OBGYN Center between 35 to 41 weeks gestation.

   Study Enrollment
2. Investigators will review charts of women scheduled for routine obstetric appointments and screen for eligibility. Eligible women will be contacted at the time of their prenatal appointment.
3. Study fliers advertising the study will also be posted in OB clinics at the OBGYN Center.
4. Women who are interested in enrollment will be counseled and consented by study personnel at their scheduled appointment.
5. The enrollment process involves a face-to-face interview with one of the study investigators for verification of study eligibility and counseling regarding study procedures as well as potential benefits and risks prior to obtaining written consent.

   Treatment Allocation
6. On day of enrollment, patients will be randomized into the treatment group or the control group using a computer-generated randomization scheme.
7. Randomization will be stratified by plan for delivery with plan for vaginal delivery versus plan for cesarean delivery, as content of the educational videos will be geared towards mode of delivery.
8. Randomization assignment will not be blinded.
9. All participants will complete an initial demographic questionnaire immediately following randomization via self- administered assessments within the test application using a mobile tablet.
10. Subjects allocated to Group 1: will:

    A. Complete the demographic questionnaire, the survey questions, and then complete the counseling aid.

    B. Prior to discharge after delivery, study personnel will administer the postpartum questionnaire via a mobile tablet. The questionnaire is programmed into the study application.
11. Subjects allocated to Group 2: will:

    A. Complete the demographic questionnaire and survey questions without watching the educational video.

    B. Prior to discharge after delivery, study personnel will administer the postpartum questionnaire via a mobile tablet. The questionnaire is programmed into the study application.
12. Research staff will complete chart reviews to confirm delivery information and other study related data.

4. Outcomes:

1. Primary: What is the impact of a standardized antepartum counseling aid on patient satisfaction with pain expectations during hospital admission for labor and delivery compared to women who do not use the counseling aid and receive routine counseling only? Satisfaction will be measured using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R). The APS-POQ-R is designed for use in adult hospital pain management QI activities and measures 6 aspects of quality including: (1) pain severity and relief; (2) impact of pain on activity, sleep, and negative emotions; (3) side effects of treatment; (4) helpfulness of information about pain treatment; (5) ability to participate in pain treatment decisions; and (6) use of nonpharmocological strategies.
2. Secondary outcomes: Perception of pain control intrapartum and postpartum based on postpartum questionnaires, expectations of what type and how much pain medication at time of discharge, use of narcotics postpartum as determined by chart review, pain perceptions in patients with history of mood disorder as determined by questionnaire, pain perceptions in patients with history of substance abuse as determined by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women > 18 years of age
2. Gestational age 35 weeks to 41 weeks
3. English or Spanish speaking
4. Plan for vaginal delivery or cesarean delivery at Greenville Memorial Hospital
5. Singleton or twin gestation

Exclusion Criteria:

1. Non-English or Non-Spanish speaking patients
2. Inability to read English, inability to read Spanish
3. Pregnancy diagnosed with fetal anomalies
4. Intrauterine fetal demise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 83 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction as measured by the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R). | 1 year
  What is the impact of a standardized antepartum counseling aid on patient satisfaction with pain expectation counseling during hospital admission for labor and delivery compared to women who do not use the counseling aid and receive routine counseling only? Satisfaction of pain expectation counseling will be measured using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R). The APS-POQ-R is designed for use in adult hospital pain management QI activities and measures 6 aspects of quality including: (1) pain severity and relief; (2) impact of pain on activity, sleep, and negative emotions; (3) side effects of treatment; (4) helpfulness of information about pain treatment; (5) ability to participate in pain treatment decisions; and (6) use of nonpharmocological strategies.
  Participants will respond on a scale of 0 to 10. 0 indicating they were extremely dissatisfied and 10 indicating they were extremely satisfied.

SECONDARY OUTCOMES:
Medication at discharge | 1 year
  Expectations of how much pain medication at time of discharge. Patient's will be asked to report what they expect to receive at discharge. Answer will be a multiple choice response. A) Tylenol/Motrin B) Narcotics 3) All of the above D) None of the above
Narcotic use | 1 year
  Amount of narcotics used in postpartum period. Charts will be reviewed to determine actual usage of narcotics during admission
Effects of pain on recovery | 1 year
  Patients will be asked how much their pain interfered with their healing or recovery. Participants will be asked to respond on a scale of 0 to 10 with 0 indicating no interference with daily activities to 10 indicating complete interference.
Pain and mood | 1 year
  Patients will be asked to rate how much their pain affected their mood. Participants will be asked to rate how much their pain affected their mood on a scale of 0 to 10 with 0 indicating not at all and 10 indicating extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Creighton Likes, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health-Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Bisch SP, Wells T, Gramlich L, Faris P, Wang X, Tran DT, Thanh NX, Glaze S, Chu P, Ghatage P, Nation J, Capstick V, Steed H, Sabourin J, Nelson G. Enhanced Recovery After Surgery (ERAS) in gynecologic oncology: System-wide implementation and audit leads to improved value and patient outcomes. Gynecol Oncol. 2018 Oct;151(1):117-123. doi: 10.1016/j.ygyno.2018.08.007. Epub 2018 Aug 9. PMID 30100053
- [Background] Scheib SA, Thomassee M, Kenner JL. Enhanced Recovery after Surgery in Gynecology: A Review of the Literature. J Minim Invasive Gynecol. 2019 Feb;26(2):327-343. doi: 10.1016/j.jmig.2018.12.010. Epub 2018 Dec 20. PMID 30580100
- [Background] Fay EE, Hitti JE, Delgado CM, Savitsky LM, Mills EB, Slater JL, Bollag LA. An enhanced recovery after surgery pathway for cesarean delivery decreases hospital stay and cost. Am J Obstet Gynecol. 2019 Oct;221(4):349.e1-349.e9. doi: 10.1016/j.ajog.2019.06.041. Epub 2019 Jun 22. PMID 31238038
- [Background] Hedderson M, Lee D, Hunt E, Lee K, Xu F, Mustille A, Galin J, Campbell C, Quesenberry C, Reyes V, Huang M, Nicol B, Paulson S, Liu V. Enhanced Recovery After Surgery to Change Process Measures and Reduce Opioid Use After Cesarean Delivery: A Quality Improvement Initiative. Obstet Gynecol. 2019 Sep;134(3):511-519. doi: 10.1097/AOG.0000000000003406. PMID 31403591
- [Background] Wilson RD, Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G. Guidelines for Antenatal and Preoperative care in Cesarean Delivery: Enhanced Recovery After Surgery Society Recommendations (Part 1). Am J Obstet Gynecol. 2018 Dec;219(6):523.e1-523.e15. doi: 10.1016/j.ajog.2018.09.015. Epub 2018 Sep 18. PMID 30240657
- [Background] Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for intraoperative care in cesarean delivery: Enhanced Recovery After Surgery Society Recommendations (Part 2). Am J Obstet Gynecol. 2018 Dec;219(6):533-544. doi: 10.1016/j.ajog.2018.08.006. Epub 2018 Aug 15. PMID 30118692
- [Background] Macones GA, Caughey AB, Wood SL, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for postoperative care in cesarean delivery: Enhanced Recovery After Surgery (ERAS) Society recommendations (part 3). Am J Obstet Gynecol. 2019 Sep;221(3):247.e1-247.e9. doi: 10.1016/j.ajog.2019.04.012. Epub 2019 Apr 14. PMID 30995461
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Peerdeman KJ, van Laarhoven AIM, Keij SM, Vase L, Rovers MM, Peters ML, Evers AWM. Relieving patients' pain with expectation interventions: a meta-analysis. Pain. 2016 Jun;157(6):1179-1191. doi: 10.1097/j.pain.0000000000000540. PMID 26945235
- [Background] Bialosky JE, Bishop MD, Cleland JA. Individual expectation: an overlooked, but pertinent, factor in the treatment of individuals experiencing musculoskeletal pain. Phys Ther. 2010 Sep;90(9):1345-55. doi: 10.2522/ptj.20090306. Epub 2010 Jun 30. PMID 20592270